CLINICAL TRIAL: NCT00354458
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Effects of KW-3902 Injectable Emulsion on Heart Failure Signs and Symptoms and Renal Function in Subjects With Acute Heart Failure Syndrome and Renal Impairment Who Are Hospitalized for Volume Overload and Require Intravenous Diuretic Therapy
Brief Title: PROTECT-2: A Study of the Selective A1 Adenosine Receptor Antagonist KW-3902 for Patients Hospitalized With Acute HF and Volume Overload to Assess Treatment Effect on Congestion and Renal Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NovaCardia, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CKI-302; 2007_804; MK7418-302
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Heart Failure, Congestive
Keywords: heart failure; diuretic; renal impairment; renal function
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — rolofylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Comparator: Placebo (unspecified)
- 2 (Experimental)
  Interventions: Drug: rolofylline

INTERVENTIONS:
Drug: rolofylline — rolofylline 30 mg IV QD; 3 days
  Other Names: KW-3902IV; MK7418
  Arms: 2
Drug: Comparator: Placebo (unspecified) — rolofylline Pbo 30 mg IV QD; 3 days
  Arms: 1

SUMMARY:
The study is being conducted to examine whether KW-3902IV will result in greater improvement in signs and symptoms of heart failure, with less treatment failure than standard therapy, when it is added to IV loop diuretics in subjects with acute heart failure syndrome and renal impairment.

DETAILED DESCRIPTION:
Loop diuretics are generally first line therapy in patients hospitalized with acute heart failure syndrome (AHFS). Their use far exceeds that of vasoactive agents. Tubuloglomerular feedback (TGF) is the body's compensatory response to avoid excess fluid loss, and it is activated when elevated sodium concentrations in the distal tubule are detected. TGF is proposed as a contributing factor for the observed diuretic resistance that occurs in patients with heart failure. Higher doses of diuretics are required to overcome the decreased natriuresis and reduced RBF induced by TGF. Ultimately, this action creates a vicious cycle of worsening renal function and diminished diuretic effectiveness.

The primary pharmacologic rationale for the use of KW-3902 in subjects with AHFS is its mechanism of action as an adenosine A1 receptor antagonist. TGF promotes release of adenosine, and adenosine binding to A1 receptors causes vasoconstriction of the afferent arteriole, decreased RBF, and enhanced sodium reabsorption by the proximal tubule. This action results in a decrease in GFR, diminished renal function, and sodium and water retention. Blocking adenosine A1 receptors via a selective adenosine receptor antagonist may limit sodium reabsorption by the proximal tubules without triggering TGF. It promotes vasodilation of the afferent arteriole of the glomerulus, and thus, this strategy offers the potential to overcome diuretic resistance or enhance diuretic responsiveness. It may also reduce the need for increasing diuretic doses that have been associated with worse outcomes.

The objectives of this study are to evaluate the effect of KW-3902IV in addition to intravenous (IV) loop diuretics (such as furosemide) on heart failure signs and symptoms, renal function, and safety in subjects hospitalized with AHFS, volume overload, and renal impairment, and to estimate and compare within-trial medical resource utilization and direct medical costs between patients treated with KW-3902IV versus placebo.

ELIGIBILITY:
Inclusion Criteria:

1. History of heart failure of at least 14 days duration for which diuretic therapy has been prescribed
2. Hospitalized for acute heart failure syndrome requiring IV diuretic therapy.
3. Impaired renal function

Exclusion Criteria:

1. Acute contrast induced nephropathy
2. Ongoing or planned IV therapy for heart failure with positive inotropic agents, vasopressors, vasodilators, or mechanical support with the exception of IV nitrates
3. BNP <500 pg/mL or NT-pro-BNP <2000 pg/mL
4. Ongoing or planned treatment with ultrafiltration, hemofiltration, or dialysis
5. Severe pulmonary disease
6. Significant stenotic valvular disease
7. Heart transplant recipient or admitted for cardiac transplantation
8. Clinical evidence of acute coronary syndrome in the 2 weeks prior to screening
9. Heart failure due to significant arrhythmias
10. Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy.
11. Known hepatic impairment
12. Non-cardiac pulmonary edema, including suspected sepsis
13. Allergy to soybean oil or eggs
14. History of seizure
15. Stroke within 2 years
16. History of or current brain tumor of any etiology
17. Brain surgery within 2 years
18. Encephalitis/meningitis within 2 years
19. History of penetrating head trauma
20. Closed head injury with loss of consciousness (LOC) over 30 minutes within 2 years
21. History of, or at risk for, alcohol withdrawal seizures
22. Advanced Alzheimer's disease
23. Advanced multiple sclerosis
24. Hgb <8 g/dL, Hct <25%, or the need for a blood transfusion
25. Previous exposure to KW-3902

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1102 (Actual)
Dates: Start 2006-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
effect on heart failure signs and symptoms | 3 Days
effect on renal function | 3 Days

SECONDARY OUTCOMES:
safety | 3 Days
within trial medical costs compared to placebo | 3 Days

CONTACTS AND LOCATIONS:
Overall Officials: Barry Massie, MD, Study Chair — University of California San Francisco, USA; Christopher O'Connor, MD, Study Chair — Duke University, USA; Marco Metra, MD, Principal Investigator — University of Brescia, Italy

REFERENCES:
- [Derived] Metra M, Cotter G, Senger S, Edwards C, Cleland JG, Ponikowski P, Cursack GC, Milo O, Teerlink JR, Givertz MM, O'Connor CM, Dittrich HC, Bloomfield DM, Voors AA, Davison BA. Prognostic Significance of Creatinine Increases During an Acute Heart Failure Admission in Patients With and Without Residual Congestion: A Post Hoc Analysis of the PROTECT Data. Circ Heart Fail. 2018 May;11(5):e004644. doi: 10.1161/CIRCHEARTFAILURE.117.004644. PMID 29748350
- [Derived] Streng KW, Ter Maaten JM, Cleland JG, O'Connor CM, Davison BA, Metra M, Givertz MM, Teerlink JR, Ponikowski P, Bloomfield DM, Dittrich HC, Hillege HL, van Veldhuisen DJ, Voors AA, van der Meer P. Associations of Body Mass Index With Laboratory and Biomarkers in Patients With Acute Heart Failure. Circ Heart Fail. 2017 Jan;10(1):e003350. doi: 10.1161/CIRCHEARTFAILURE.116.003350. PMID 28069685
- [Derived] Matsue Y, van der Meer P, Damman K, Metra M, O'Connor CM, Ponikowski P, Teerlink JR, Cotter G, Davison B, Cleland JG, Givertz MM, Bloomfield DM, Dittrich HC, Gansevoort RT, Bakker SJ, van der Harst P, Hillege HL, van Veldhuisen DJ, Voors AA. Blood urea nitrogen-to-creatinine ratio in the general population and in patients with acute heart failure. Heart. 2017 Mar;103(6):407-413. doi: 10.1136/heartjnl-2016-310112. Epub 2016 Sep 22. PMID 27658757
- [Derived] Ter Maaten JM, Damman K, Hanberg JS, Givertz MM, Metra M, O'Connor CM, Teerlink JR, Ponikowski P, Cotter G, Davison B, Cleland JG, Bloomfield DM, Hillege HL, van Veldhuisen DJ, Voors AA, Testani JM. Hypochloremia, Diuretic Resistance, and Outcome in Patients With Acute Heart Failure. Circ Heart Fail. 2016 Aug;9(8):e003109. doi: 10.1161/CIRCHEARTFAILURE.116.003109. PMID 27507112
- [Derived] Tromp J, Meyer S, Mentz RJ, O'Connor CM, Metra M, Dittrich HC, Ponikowski P, Teerlink JR, Cotter G, Davison B, Cleland JG, Givertz MM, Bloomfield DM, van Veldhuisen DJ, Hillege HL, Voors AA, van der Meer P. Acute heart failure in the young: Clinical characteristics and biomarker profiles. Int J Cardiol. 2016 Oct 15;221:1067-72. doi: 10.1016/j.ijcard.2016.06.339. Epub 2016 Jul 5. PMID 27448534
- [Derived] Ter Maaten JM, Valente MA, Damman K, Cleland JG, Givertz MM, Metra M, O'Connor CM, Teerlink JR, Ponikowski P, Bloomfield DM, Cotter G, Davison B, Subacius H, van Veldhuisen DJ, van der Meer P, Hillege HL, Gheorghiade M, Voors AA. Combining Diuretic Response and Hemoconcentration to Predict Rehospitalization After Admission for Acute Heart Failure. Circ Heart Fail. 2016 Jun;9(6):e002845. doi: 10.1161/CIRCHEARTFAILURE.115.002845. PMID 27266853
- [Derived] Givertz MM, Postmus D, Hillege HL, Mansoor GA, Massie BM, Davison BA, Ponikowski P, Metra M, Teerlink JR, Cleland JG, Dittrich HC, O'Connor CM, Cotter G, Voors AA. Renal function trajectories and clinical outcomes in acute heart failure. Circ Heart Fail. 2014 Jan;7(1):59-67. doi: 10.1161/CIRCHEARTFAILURE.113.000556. Epub 2013 Nov 26. PMID 24281137
- [Derived] Cleland JG, Chiswell K, Teerlink JR, Stevens S, Fiuzat M, Givertz MM, Davison BA, Mansoor GA, Ponikowski P, Voors AA, Cotter G, Metra M, Massie BM, O'Connor CM. Predictors of postdischarge outcomes from information acquired shortly after admission for acute heart failure: a report from the Placebo-Controlled Randomized Study of the Selective A1 Adenosine Receptor Antagonist Rolofylline for Patients Hospitalized With Acute Decompensated Heart Failure and Volume Overload to Assess Treatment Effect on Congestion and Renal Function (PROTECT) Study. Circ Heart Fail. 2014 Jan;7(1):76-87. doi: 10.1161/CIRCHEARTFAILURE.113.000284. Epub 2013 Nov 26. PMID 24281134
- [Derived] Teerlink JR, Iragui VJ, Mohr JP, Carson PE, Hauptman PJ, Lovett DH, Miller AB, Pina IL, Thomson S, Varosy PD, Zile MR, Cleland JG, Givertz MM, Metra M, Ponikowski P, Voors AA, Davison BA, Cotter G, Wolko D, Delucca P, Salerno CM, Mansoor GA, Dittrich H, O'Connor CM, Massie BM. The safety of an adenosine A(1)-receptor antagonist, rolofylline, in patients with acute heart failure and renal impairment: findings from PROTECT. Drug Saf. 2012 Mar 1;35(3):233-44. doi: 10.2165/11594680-000000000-00000. PMID 22339573
- [Derived] O'Connor CM, Fiuzat M, Lombardi C, Fujita K, Jia G, Davison BA, Cleland J, Bloomfield D, Dittrich HC, Delucca P, Givertz MM, Mansoor G, Ponikowski P, Teerlink JR, Voors AA, Massie BM, Cotter G, Metra M. Impact of serial troponin release on outcomes in patients with acute heart failure: analysis from the PROTECT pilot study. Circ Heart Fail. 2011 Nov;4(6):724-32. doi: 10.1161/CIRCHEARTFAILURE.111.961581. Epub 2011 Sep 6. PMID 21900185
- [Derived] Voors AA, Dittrich HC, Massie BM, DeLucca P, Mansoor GA, Metra M, Cotter G, Weatherley BD, Ponikowski P, Teerlink JR, Cleland JG, O'Connor CM, Givertz MM. Effects of the adenosine A1 receptor antagonist rolofylline on renal function in patients with acute heart failure and renal dysfunction: results from PROTECT (Placebo-Controlled Randomized Study of the Selective Adenosine A1 Receptor Antagonist Rolofylline for Patients Hospitalized with Acute Decompensated Heart Failure and Volume Overload to Assess Treatment Effect on Congestion and Renal Function). J Am Coll Cardiol. 2011 May 10;57(19):1899-907. doi: 10.1016/j.jacc.2010.11.057. PMID 21545947
- [Derived] Massie BM, O'Connor CM, Metra M, Ponikowski P, Teerlink JR, Cotter G, Weatherley BD, Cleland JG, Givertz MM, Voors A, DeLucca P, Mansoor GA, Salerno CM, Bloomfield DM, Dittrich HC; PROTECT Investigators and Committees. Rolofylline, an adenosine A1-receptor antagonist, in acute heart failure. N Engl J Med. 2010 Oct 7;363(15):1419-28. doi: 10.1056/NEJMoa0912613. PMID 20925544
- [Derived] Cotter G, Dittrich HC, Weatherley BD, Bloomfield DM, O'Connor CM, Metra M, Massie BM; Protect Steering Committee, Investigators, and Coordinators. The PROTECT pilot study: a randomized, placebo-controlled, dose-finding study of the adenosine A1 receptor antagonist rolofylline in patients with acute heart failure and renal impairment. J Card Fail. 2008 Oct;14(8):631-40. doi: 10.1016/j.cardfail.2008.08.010. Epub 2008 Sep 14. PMID 18926433